CLINICAL TRIAL: NCT00483561
Title: A Phase II Study Evaluating the Efficacy of Iressa Plus Etoposide in Patients With Advanced Hormone Refractory Prostate Cancer
Brief Title: Gefitinib and Etoposide in Treating Patients With Advanced Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left UNMC
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0285-03-FB; P30CA036727 (NIH)
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gefitinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gefitinib plus Etoposide (Experimental): Gefitinib 250 mg p.o. daily, starting on Day 1and taken on a continuous basis throughout the trial.
  Etoposide 50 mg/m2/day for Days 1-14 out of a 28-day cycle. (Etoposide capsules come in a 50-mg dose formulation, and the patient's dose will be rounded to the nearest 50-mg multiple).
  Interventions: Drug: Gefitinib plus etoposide

INTERVENTIONS:
Drug: Gefitinib plus etoposide — Gefitinib 250 mg p.o. daily, starting on Day 1and taken on a continuous basis throughout the trial with Etoposide 50 mg/m2/day for Days 1-14 out of a 28-day cycle. (Etoposide capsules come in a 50-mg dose formulation, and the patient's dose will be rounded to the nearest 50-mg multiple).
  Other Names: Iressa; ZD1839

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gefitinib together with etoposide may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gefitinib together with etoposide works in treating patients with advanced prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity of gefitinib and etoposide, in terms of overall response rate, in patients with hormone-refractory advanced prostate cancer previously treated with docetaxel-based therapy.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine whether related biomarkers can help predict response in patients treated with this regimen.

OUTLINE: This is a nonrandomized study.

Patients receive oral gefitinib once daily on days 1-28 and oral etoposide once daily on days 1-14. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and periodically during study for correlative studies. Blood samples are analyzed by enzyme-linked immunosorbent assays for biomarkers (e.g., VEGF, basic fibroblast growth factor, and anti-EGFR antibody titers) in order to determine whether one or more of these biomarkers can predict response.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Progressive disease after a prior docetaxel-based regimen OR failed a prior docetaxel-based regimen
* Hormone-refractory disease, meeting 1 of the following criteria:
* Radiologically measurable disease
* Prostate-specific antigen (PSA) progression* while on hormonal therapy (including withdrawal from a direct antagonist) NOTE: *If the confirmatory PSA value is less than the screening PSA value, then an additional test for rising PSA is required to document progression
* Must have undergone prior surgical castration OR currently be on a luteinizing hormone-releasing hormone agonistANC > 1,500/mm³Platelet count > 100,000/mm³Hemoglobin > 10 g/dL (in the absence of packed red blood cell transfusions within the past 4 weeks)Creatinine < 2 mg/dLAST and ALT < 2 times upper limit of normal (ULN)Alkaline phosphatase < 2 times ULNFertile patients must use effective double-method contraception during and for 1 month after completion of study treatmentAt least 4 weeks since prior cytotoxic therapy
* At least 4 weeks since prior direct antagonists, including flutamide and nilutamide
* At least 6 weeks since prior bicalutamide
* At least 30 days since prior nonapproved or investigational drugs
* More than 4 weeks since prior palliative radiotherapy o The irradiated lesion must not be used to assess response rate

Exclusion Criteria:

* No other malignancy within the past 5 years except basal cell carcinoma
* No clinically significant New York Heart Association class II-IV cardiovascular disease
* No evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* No unresolved chronic toxicity > grade 2 from prior anticancer therapy, with the exception of alopecia
* No other significant clinical disorder or laboratory finding that would preclude study participation
* No known severe hypersensitivity to gefitinib or any of the excipients of this product
* No evidence of clinically active interstitial lung disease

  o Asymptomatic Patients with chronic, stable radiographic changes are eligible
* No prior gefitinib or etoposide
* No concurrent palliative radiotherapy
* No concurrent chemotherapeutic agents
* No concurrent phenytoin, carbamazepine, rifampin, barbiturates, or Hypericum perforatum (St. John's wort)
* No concurrent hormones except antiandrogen therapy, steroids for adrenal failure, hormones for nondisease-related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic
* No concurrent initiation of IV and/or oral bisphosphonates specifically for symptomatic bone metastases

Ages: 19 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hauke, MD, Principal Investigator — University of Nebraska; Elizabeth C Reed, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gefitinib Plus Etoposide: Gefitinib plus etoposide: Gefitinib 250 mg p.o. daily, starting on Day 1 and taken on a continuous basis throughout the trial with Etoposide-50 mg/m2/day for Days 1-14 out of a 28-day cycle. (Etoposide capsules come in a 50-mg dose formulation, and the patient's dose will be rounded to the nearest 50-mg multiple).
  Patients with stable disease will be treated for 2 additional cycles beyond maximum response, for a maximum of 6 cycles. Restaging will be performed every 2 cycles. After completion of treatment, patients will continue to be followed for survival.
Period: Overall Study
Arm/Group | Gefitinib Plus Etoposide
Started | 26
Completed | 15
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Gefitinib Plus Etoposide
Number analyzed (Participants) | 26
Age, Customized [Count of Participants; unit: Participants]
  Number of subjects 19 years of age and older | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate as Measured by RECIST Criteria and PSA Criteria
Description: If there is at least 1 response, then 7 additional patients will be enrolled. If there are 4 or more responders overall, then the combination will be considered active and warrant further study. Overall response rate (ORR) is defined as the proportion of patients who have a partial or complete response to therapy.
Time Frame: Approximately 3 years
Population: Fifteen subjects were evaluable. A total of 26 subjects were consented; two were screen failures. Nine subjects were not evaluable due to coming off study prior to reaching the point of evaluation (2 cycles).
Measure: Count of Participants; unit: Participants
Arm/Group | Gefitinib Plus Etoposide
Number analyzed (Participants) | 15
Participants
  Stable Disease (by RECIST criteria) | 5
  Partial Responder (by PSA criteria) | 1

2. Secondary Outcome: Biomarkers
Time Frame: At every cycle
Population: Evaluation of this data is not possible as the investigator performing the analysis has left the study center prior to completing the analysis and data was not provided.
Arm/Group | Gefitinib Plus Etoposide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 52 months
Groups:
- Gefitinib Plus Etoposide: Gefitinib 250 mg p.o. daily, starting on Day 1and taken on a continuous basis throughout the trial.
  Etoposide 50 mg/m2/day for Days 1-14 out of a 28-day cycle. (Etoposide capsules come in a 50-mg dose formulation, and the patient's dose will be rounded to the nearest 50-mg multiple).
  Gefitinib plus etoposide: Gefitinib 250 mg p.o. daily, starting on Day 1and taken on a continuous basis throughout the trial with Etoposide 50 mg/m2/day for Days 1-14 out of a 28-day cycle. (Etoposide capsules come in a 50-mg dose formulation, and the patient's dose will be rounded to the nearest 50-mg multiple).
Arm/Group | Gefitinib Plus Etoposide
All-Cause Mortality (participants affected / at risk) | 14/26
Serious Adverse Events (participants affected / at risk) | 7/26
Other Adverse Events (participants affected / at risk) | 4/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib Plus Etoposide (N=26)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) — Pulmonary embolism
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) — Hemoglobin
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — shortness of breath
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) — deep vein thrombosis
Seizure (Nervous system disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Acute renal failure
Hypotension (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — weakness
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib Plus Etoposide (N=26)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 (5) — hemoglobin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No